CLINICAL TRIAL: NCT01415518
Title: Efficacy and Tolerability Study of Symbicort Turbuhaler(160/4.5µg/Inhalation,2inhalations Twice Daily) Added to Atrovent (20µg/Inhalation, 2 Inhalations 4 Times Daily)+Theophylline SR(0.1g/Tablet,1 Tablet p.o. Twice Daily) Compared With Atrovent+Theophylline SR in Severe COPD Patients.
Brief Title: Efficacy and Tolerability Study in Severe Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: SECURE2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D589BL00022
Record Dates: First submitted 2011-08-08; First posted 2011-08-12 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2019-07-09 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Severe chronic obstructive pulmonary disease (COPD) patients
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Budesonide; Formoterol Fumarate; Budesonide, Formoterol Fumarate Drug Combination; Ipratropium; Theophylline

ARMS (2):
- 1 (Other): budesonide/formoterol (Symbicort Turbuhaler 160/4.5µg/inhalation, 2 inhalations twice daily) added to ipratropium (AtroventTM 20 µg/inhalation, 2 inhalations four times daily) + theophylline SR (0.1g/tablet, 1 tablet p.o. twice daily)
  Interventions: Drug: Drug: Budesonide/formoterol (Symbicort Turbuhaler; Drug: Drug: ipratropium (AtroventTM); Drug: theophylline SR
- 2 (Other): ipratropium (AtroventTM 20 µg/inhalation, 2 inhalations four times daily) + theophylline SR (0.1g/tablet, 1 tablet p.o. twice daily)
  Interventions: Drug: Drug: ipratropium (AtroventTM); Drug: theophylline SR

INTERVENTIONS:
Drug: Drug: Budesonide/formoterol (Symbicort Turbuhaler — budesonide/formoterol (Symbicort Turbuhaler 160/4.5µg/inhalation, 2 inhalations twice daily)
  Arms: 1
Drug: Drug: ipratropium (AtroventTM) — ipratropium (AtroventTM 20 µg/inhalation, 2 inhalations four times daily)
Drug: theophylline SR — theophylline SR (0.1g/tablet, 1 tablet p.o. twice daily)

SUMMARY:
Efficacy and tolerability study in severe chronic obstructive pulmonary disease (COPD) patients.

DETAILED DESCRIPTION:
Efficacy and tolerability study of Symbicort Turbuhaler (160/4.5µg/inhalation,2inhalations twice daily) added to Atrovent (20µg/inhalation, 2 inhalations 4 times daily) + theophylline SR(0.1g/tablet, 1 tablet p.o. twice daily) compared with Atrovent + theophylline SR in severe COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent
* Men or women patients ≥ 40 years of age
* Diagnosis of COPD with symptoms for more than 2 years and there is a history of at least one COPD exacerbation requiring a course of oral steroids and/or antibiotics within 1-12 months before Visit 2
* Forced Expiratory Volume in 1 second (FEV1) ≤50% of predicted normal value, pre-bronchodilator and Forced Expiratory Volume in 1 second (FEV1) / Forced Vital Capacity (FVC) < 70%, pre-bronchodilator
* Total symptom score of 2 or more per day for at least half of run-in period (breathing, cough and sputum scores from the diary card) and complete morning recordings of Digital Peak Flow Meter data at least 7 out of the last 10 days of the run-in period

Exclusion Criteria:

* A history of asthma and seasonal allergic rhinitis before 40 years of age
* Patients who have experienced exacerbation of COPD requiring hospitalisation and /or emergency room treatment and/or a course of oral steroids and/or intravenous corticosteroids and/or antibiotics within 4 weeks prior to Visit 2 and/or during run-in period
* Patients with relevant cardiovascular disorder judged by the investigator
* Patients with glaucoma, prostatic hyperplasia or bladder-neck obstruction judged by the investigator
* Women who are pregnant, breast-feeding or of child-bearing potential judged by the investigator

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 581 (Actual)
Dates: Start 2011-09-01 (Actual); Primary Completion 2012-12-01 (Actual); Study Completion 2012-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Chen, Study Chair — AstraZeneca Singapore Pte Ltd
Locations (21):
- China (21):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Foshan, Guangdong
  - Research Site, Guangzhou, Guangdong
  - Research Site, Zhongshan, Guangdong
  - Research Site, Haikou, Hainan
  - Research Site, Shijiazhuang, Hebei
  - Research Site, Tangshan, Hebei
  - Research Site, Zhengzhou, Henan
  - Research Site, Wuhan, Hubei
  - Research Site, Changsha, Hunan
  - Research Site, Nanjing, Jiangsu
  - Research Site, Changchun, Jilin
  - Research Site, Shenyang, Liaoning
  - Research Site, Qingdao, Shandong
  - Research Site, Shanghai, Shanghai Municipality
  - Research Site, Tianjin, Tianjin Municipality
  - Research Site, Chengdu
  - Research Site, Chongqin
  - Research Site, Dalian
  - Research Site, Ha'er BING
  - Research Site, Hohhot

REFERENCES:
- See also: Clinical Study Protocol — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D589BL00022&attachmentIdentifier=2a7ff667-339c-456d-8acc-8e6f547b9c3d&fileName=D589BL00022_Clinical_Study_Protocol_REDACTED.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D589BL00022&attachmentIdentifier=816840bb-da84-40c7-b174-fa5951b2c915&fileName=D589BL00022_SECURE2_Synopsis_1_0_20131126_v2.0001-v4.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Groups:
- Symbicort Turbuhaler + Ipratropium + Theophylline SR: Symbicort Turbuhaler 160/4.5μg/inhalation, 2 inhalations twice daily) added to ipratropium (AtroventTM 20 μg/inhalation, 2 inhalations four times daily) + theophylline SR (0.1g/tablet, 1 tablet p.o. twice daily)
- Ipratropium + Theophylline SR: ipratropium (AtroventTM 20 μg/inhalation, 2 inhalations four times daily) + theophylline SR (0.1g/tablet, 1 tablet p.o. twice daily)
Period: Overall Study
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Started | 292 | 292
Patients Who Received Study Treatment | 290 | 292
Pts With Correct Randomized Treatment | 290 (Efficacy analysis used 290 patients. Safety analysis used 290+3=293 patients.) | 289 (Efficacy analysis used 292 patients. Safety analysis used 292-3=289 patients.)
Completed | 276 | 261
Not Completed | 16 | 31
Not completed — Withdrawal by Subject | 2 | 12
Not completed — Protocol Violation | 6 | 8
Not completed — Lost to Follow-up | 3 | 5
Not completed — Adverse Event | 3 | 4
Not completed — Death | 1 | 1
Not completed — Condition under Investigation Worsened | 1 | 1

BASELINE CHARACTERISTICS:
Population: Two patients in 'Symbicort Turbuhaler + ipratropium + theophylline' group did not receive study treatment and were excluded from the analysis popolation. Thus the number of patients in that group is 290 (= 290 - 2).
Groups:
- Total: Total of all reporting groups
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR | Total
Number analyzed (Participants) | 290 | 292 | 582
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (8.79) | 64.4 (8.76) | 64.1 (8.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 43 | 79
  Male | 254 | 249 | 503

OUTCOME MEASURES:

1. Primary Outcome: Pre-dose FEV1
Description: Ratio of pre-dose FEV1 (Forced Expiratory Volume in 1 second) in treatment period to baseline value
Time Frame: Baseline (week 0) and mean in treatment period (weeks 1, 6, 12) measured before inhalation of study drug
Population: FAS
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 286 | 286
Ratio | 1.079 [1.059 to 1.100] | 1.009 [0.990 to 1.029]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p < .0001, ANCOVA; multiplicative ANCOVA model with treatment and centre as fixed factors and baseline value as a (log-transformed) covariate; Ratio = 1.069, 95% CI 2-sided [1.043 to 1.096]

2. Secondary Outcome: Post-dose FEV1 at 5 Minutes
Description: Ratio of post-dose FEV1 at 5 minutes to baseline value
Time Frame: Baseline (-2 weeks) and mean in treatment period (1, 6, 12 weeks) measured at 5 minutes after inhalation of study drug
Population: FAS
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 288 | 292
Ratio | 1.179 [1.161 to 1.199] | 1.106 [1.088 to 1.124]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio = 1.067, 95% CI 2-sided [1.044 to 1.090]

3. Secondary Outcome: Post-dose FEV1 at 60 Minutes
Description: Ratio of post-dose FEV1 at 60 minutes to baseline value
Time Frame: Baseline (meaured before inhalation of study drug at week 0) and mean in treatment period (measured at 1 hour after inhalation of study drug at weeks 0, 1, 6, 12)
Population: FAS
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 288 | 292
Ratio | 1.219 [1.199 to 1.240] | 1.142 [1.123 to 1.162]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio = 1.068, 95% CI [1.043 to 1.092]

4. Secondary Outcome: Pre-dose FVC
Description: Ratio of pre-dose FVC (Forced Vital Capacity) to baseline
Time Frame: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 286 | 286
Ratio | 1.072 [1.054 to 1.090] | 1.030 [1.013 to 1.048]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0007, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio = 1.040, 95% CI 2-sided [1.017 to 1.064]

5. Secondary Outcome: Post-dose FVC at 5 Minutes
Description: Ratio of post-dose FVC at 5 minutes to baseline
Time Frame: Baseline (meaured before inhalation of study drug at week 0) and mean in treatment period (measured at 5 minutes after inhalation of study drug at weeks 0, 1, 6, 12)
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 288 | 292
Ratio | 1.170 [1.153 to 1.188] | 1.120 [1.104 to 1.137]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p < .0001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio = 1.045, 95% CI 2-sided [1.024 to 1.065]

6. Secondary Outcome: Post-dose FVC at 60 Minutes
Description: Ratio of post-dose FVC at 60 minutes to baseline
Time Frame: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 288 | 292
Ratio | 1.192 [1.174 to 1.211] | 1.148 [1.130 to 1.166]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0003, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio = 1.038, 95% CI 2-sided [1.017 to 1.060]

7. Secondary Outcome: Pre-dose IC
Description: Ratio of pre-dose IC (Inspiratory Capacity) to baseline
Time Frame: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 276 | 264
Ratio | 1.068 [1.045 to 1.092] | 1.032 [1.010 to 1.056]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0248, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio = 1.035, 95% CI 2-sided [1.004 to 1.066]

8. Secondary Outcome: Post-dose IC at 60 Minutes
Description: Ratio of post-dose IC at 60 minutes to baseline
Time Frame: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 278 | 271
Ratio | 1.163 [1.140 to 1.187] | 1.120 [1.097 to 1.143]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0074, ANCOVA; [statistical method as in outcome 1, analysis 1]; Ratio = 1.038, 95% CI 2-sided [1.010 to 1.067]

9. Secondary Outcome: Pre-dose PEF in Last Week of Treatment
Description: Change in pre-dose morning PEF (Peak Expiratory Flow) from run-in period to last week of treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured before inhalation of study drug in the last week of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 207 | 191
L/min | 23.135 [13.808 to 32.462] | -2.038 [-11.678 to 7.603]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0001, ANCOVA; Additive ANCOVA model with treatment and centre as fixed factors and the run-in mean of pre-dose morning PEF as a covariate; Mean Difference (Net) = 25.172, 95% CI 2-sided [12.733 to 37.611]

10. Secondary Outcome: Pre-dose PEF in First Week of Treatment
Description: Change in pre-dose morning PEF from run-in period to first week of treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurments measured before inhalation of study drug in the first week of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 228 | 215
L/min | 24.393 [16.799 to 31.987] | 3.257 [-4.357 to 10.871]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p < .0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 21.136, 95% CI 2-sided [12.163 to 30.110]

11. Secondary Outcome: Pre-dose PEF in Whole Treatment Period
Description: Change in pre-dose morning PEF from run-in period to whole treatment period
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured before inhalation of study drug in whole treatment period (12 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 247 | 246
L/min | 21.021 [14.563 to 27.479] | -2.023 [-8.555 to 4.510]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p < .0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 23.044, 95% CI 2-sided [14.927 to 31.161]

12. Secondary Outcome: Post-dose PEF in Last Week of Treatment
Description: Change in post-dose morning PEF at 5 minutes from run-period to last week of treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured at 5 minutes after inhalation of study drug in the last week of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 158 | 156
L/min | 36.612 [26.656 to 46.569] | 5.100 [-4.702 to 14.901]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p < .0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 31.513, 95% CI 2-sided [18.740 to 44.286]

13. Secondary Outcome: Post-dose PEF in First Week of Treatment
Description: Change in post-dose morning PEF at 5 minutes from run-in period to first week of treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurments measured at 5 minutes after inhalation of study drug in the first week of treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 170 | 179
L/min | 25.993 [17.330 to 34.656] | 1.670 [-6.582 to 9.922]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p < .0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 24.322, 95% CI 2-sided [14.425 to 34.220]

14. Secondary Outcome: Post-dose PEF in Whole Treatment Period
Description: Change in post-dose morning PEF at 5 minutes from run-period to whole treatment period
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured at 5 minutes after inhalation of study drug in whole treatment period (12 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: L/min
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 237 | 239
L/min | 26.507 [19.892 to 33.122] | -0.662 [-7.278 to 5.955]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p < .0001, ANCOVA; [statistical method as in outcome 9, analysis 1]; Mean Difference (Net) = 27.168, 95% CI 2-sided [18.906 to 35.431]

15. Secondary Outcome: Use of Reliever Medication During Day in the Last Week on Treatment
Description: Change in the number of inhalations of reliever medication during day from run-in to the last week on treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured during day in the last week on treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: times/day
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 273 | 266
times/day | -0.398 [-0.570 to -0.226] | -0.101 [-0.276 to 0.074]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0102, ANCOVA; Additive ANCOVA model with treatment and centre as fixed factors and the run-in mean of reliever medication as a covariate; Mean Difference (Net) = -0.297, 95% CI 2-sided [-0.522 to -0.071]

16. Secondary Outcome: Use of Reliever Medication During Day in the First Week on Treatment
Description: Change in the number of inhalations of reliever medication during day from run-in to the first week on treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured during day in the first week on treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: times/day
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 283 | 282
times/day | -0.440 [-0.583 to -0.297] | -0.097 [-0.241 to 0.047]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0004, ANCOVA; [statistical method as in outcome 15, analysis 1]; Mean Difference (Net) = -0.343, 95% CI 2-sided [-0.533 to -0.153]

17. Secondary Outcome: Use of Reliever Medication During Day in the Whole Treatment Period
Description: Change in the number of inhalations of reliever medication during day from run-in to the whole treatment period
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured during day in the whole treatment period (12 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: times/day
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 283 | 285
times/day | -0.404 [-0.539 to -0.268] | -0.061 [-0.197 to 0.075]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0002, ANCOVA; [statistical method as in outcome 15, analysis 1]; Mean Difference (Net) = -0.342, 95% CI 2-sided [-0.523 to -0.162]

18. Secondary Outcome: Change in COPD Symptoms - Breathing
Description: Change in breathing symptom score (from 0 (none) to 4 (severe)) from run-in period
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements in the whole treatment period (12 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: Score from 0 to 4
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 284 | 287
Score from 0 to 4 | -0.507 [-0.584 to -0.431] | -0.229 [-0.305 to -0.152]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p < .0001, ANCOVA; Additive ANCOVA model with treatment and centre as fixed factors and the run-in mean of score as a covariate; Mean Difference (Net) = -0.279, 95% CI 2-sided [-0.381 to -0.177]

19. Secondary Outcome: COPD Symptoms - Cough
Description: Change in cough symptom score (from 0 (none) to 4 (almost constant)) from run-in period
Time Frame: as for outcome 18
Measure: Least Squares Mean (95% Confidence Interval); unit: Score from 0 to 4
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 284 | 287
Score from 0 to 4 | -0.441 [-0.516 to -0.365] | -0.248 [-0.324 to -0.172]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0002, ANCOVA; Additive ANCOVA model with treatment and centre as fixed factors and the run-in mean of score as a covariate; Mean Difference (Net) = -0.193, 95% CI 2-sided [-0.294 to -0.092]

20. Secondary Outcome: COPD Symptoms Sputum
Description: Change in sputum symptom score (from 0 (none) to 4 (severe)) from run-in period
Time Frame: as for outcome 18
Measure: Least Squares Mean (95% Confidence Interval); unit: Score from 0 to 4
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 284 | 287
Score from 0 to 4 | -0.332 [-0.407 to -0.257] | -0.124 [-0.200 to -0.049]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0001, ANCOVA; Additive ANCOVA model with treatment and centre as fixed factors and the run-in mean of score as a covariate; Mean Difference (Net) = -0.208, 95% CI 2-sided [-0.308 to -0.108]

21. Secondary Outcome: COPD Exacerbations
Description: Severe exacerbations requiring systemic steroids (oral ≥3 days or parenteral) or hospitalisation or emergency room treatment due to worsening of COPD symptoms
Time Frame: Whole treatment period (12 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: exacerbations/12 weeks
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 290 | 292
exacerbations/12 weeks | 0.069 [0.044 to 0.106] | 0.121 [0.087 to 0.170]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0425, Poisson regression; Poisson regression model with treatment as a factor and the duration time in study as an offset variable; Rate ratio = 0.565, 95% CI 2-sided [0.325 to 0.981]
Statistical Analysis 2: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0880, Regression, Cox; Time to the first COPD exacerbation; Hazard Ratio (HR) = 0.604, 95% CI 2-sided [0.339 to 1.078]
Statistical Analysis 3: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0845, Log Rank; Time to the first COPD exacerbation

22. Secondary Outcome: Use of Reliever Medication During Night in the Last Week on Treatment
Description: Change in the number of inhalations of reliever medication during day from run-in to the whole treatment period
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured during night in the last week on treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: times/day
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 269 | 263
times/day | -0.078 [-0.147 to -0.009] | -0.023 [-0.093 to 0.046]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.2281, ANCOVA; [statistical method as in outcome 15, analysis 1]; Mean Difference (Net) = -0.055, 95% CI 2-sided [-0.144 to 0.035]

23. Secondary Outcome: Use of Reliever Medication During Night in the First Week on Treatment
Description: change in the number of inhalations of reliever medication during day from run-in to the first week on treatment
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured during night in the first week on treatment
Measure: Least Squares Mean (95% Confidence Interval); unit: times/day
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 278 | 282
times/day | -0.124 [-0.179 to -0.068] | -0.002 [-0.057 to 0.053]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0010, ANCOVA; [statistical method as in outcome 15, analysis 1]; Mean Difference (Net) = -0.122, 95% CI 2-sided [-0.194 to -0.049]

24. Secondary Outcome: Use of Reliever Medication During Night in the Whole Treatment Period
Description: Change in the number of inhalations of reliever medication during day from run-in to the whole treatment period
Time Frame: Mean of daily measurements in run-in period (the last 10 days before randomization) and mean of daily measurements measured during night in the whole treatment period (12 weeks)
Measure: Least Squares Mean (95% Confidence Interval); unit: times/day
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Number analyzed (Participants) | 280 | 284
times/day | -0.086 [-0.144 to -0.027] | 0.020 [-0.038 to 0.079]
Statistical Analysis 1: Comparison: Symbicort Turbuhaler + Ipratropium + Theophylline SR vs Ipratropium + Theophylline SR; Test type: Superiority or Other; p = 0.0073, ANCOVA; [statistical method as in outcome 15, analysis 1]; Mean Difference (Net) = -0.106, 95% CI 2-sided [-0.183 to -0.029]

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Symbicort Turbuhaler + Ipratropium + Theophylline SR | Ipratropium + Theophylline SR
Serious Adverse Events (participants affected / at risk) | 9/293 | 10/289
Other Adverse Events (participants affected / at risk) | 33/293 | 31/289
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort Turbuhaler + Ipratropium + Theophylline SR (N=293) | Ipratropium + Theophylline SR (N=289)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Fungal oesophagitis (Gastrointestinal disorders) | 1 | 0
Gastritis atrophic (Gastrointestinal disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Erysipelas (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Symbicort Turbuhaler + Ipratropium + Theophylline SR (N=293) | Ipratropium + Theophylline SR (N=289)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 7
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pyrexia (General disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Dizziness (Nervous system disorders) | 1 | 1
Palpitations (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Fungal oesophagitis (Gastrointestinal disorders) | 1 | 0
Gastritis atrophic (Gastrointestinal disorders) | 1 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Chest discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asphyxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infection (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chest discomfort (General disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint sprain (Injury, poisoning and procedural complications) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 1
Erysipelas (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema of eyelid (Skin and subcutaneous tissue disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall not publish any results until the earlier of (i) the date of the first Study results publication authorized by AZ and (ii) the end of the 18 month period following the completion of the Study. PI shall provide AZ with such material for review, at least 60 days prior to submission for publication. If requested in writing by AZ, PI shall withhold material from submission for publication for an additional 90 days from the date of AZ's request.